CLINICAL TRIAL: NCT02615262
Title: Intraoperative Dexamethasone in Pediatric Cardiac Surgery: a Prospective Double-blind Randomised Clinical Trial
Brief Title: Intraoperative Dexamethasone in Pediatric Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dex01
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Cardiac Surgery; Congenital Heart Defects; Cardiopulmonary Bypass
Keywords: Pediatric cardiac surgery; Dexamethasone; Steroids; Cardiopulmonary bypass; Congenital heart defects; Infants
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Dexamethasone 1 mg per 1 kg of body weight intravenously immediately after induction of anesthesia
  Interventions: Drug: Dexamethasone
- Control (Placebo Comparator): 0.9% Sodium Chloride 0.25 ml per 1 kg of body weight intravenously immediately after induction of anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Experimental
Drug: Placebo — 0.9% Sodium Chloride
  Arms: Control

SUMMARY:
Perioperative administration of steroids has been demonstrated to reduce systemic inflammatory response in infants undergoing cardiac surgery with cardiopulmonary bypass. However, data on effects of steroids on clinical outcomes are lacking. Hence the hypothesis of the present study: intraoperative administration of dexamethasone reduces complication rates and improves clinical outcomes in infants undergoing repair of congenital heart defects under cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* elective repair of congenital heart defects under cardiopulmonary bypass

Exclusion Criteria:

* absence of written informed consent signed by parent or guardian;
* hypoplastic left heart syndrome;
* participation in conflicting randomised studies;
* emergency surgery;
* inotropic support prior to surgery;
* mechanical ventilation prior to surgery;
* bacterial, viral or fungal infection in the preceding 30 days;
* gestational age less that 37 weeks;
* perinatal central nervous system damage.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 394 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Major complications | 30 days after surgery
  Composite of all-cause death, myocardial infarction, need for extracorporeal membrane oxygenation implantation, cardiac arrest, acute renal failure (stage "injury" or higher according to pRIFLE scale), prolonged mechanical ventilation (> 24 hours), stroke, seizure, coma.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lomivorotov, PhD, Principal Investigator — Novosibirsk Research Institute of Circulation Pathology
Locations (4):
- Dante Pazzanese Cardiology Institute, São Paulo, Brazil
- Shanghai Childrens Medical Center, Shanghai, China
- Russia (2):
  - Novosibirsk Research Institute of Circulation Pathology, Novosibirsk
  - Federal Center of Cardiovascular Surgery, Penza city, Penza

REFERENCES:
- [Derived] Gibbison B, Villalobos Lizardi JC, Aviles Martinez KI, Fudulu DP, Medina Andrade MA, Perez-Gaxiola G, Schadenberg AW, Stoica SC, Lightman SL, Angelini GD, Reeves BC. Prophylactic corticosteroids for paediatric heart surgery with cardiopulmonary bypass. Cochrane Database Syst Rev. 2020 Oct 12;10(10):CD013101. doi: 10.1002/14651858.CD013101.pub2. PMID 33045104
- [Derived] Lomivorotov V, Kornilov I, Boboshko V, Shmyrev V, Bondarenko I, Soynov I, Voytov A, Polyanskih S, Strunin O, Bogachev-Prokophiev A, Landoni G, Nigro Neto C, Oliveira Nicolau G, Saurith Izquierdo L, Nogueira Nascimento V, Wen Z, Renjie H, Haibo Z, Bazylev V, Evdokimov M, Sulejmanov S, Chernogrivov A, Ponomarev D. Effect of Intraoperative Dexamethasone on Major Complications and Mortality Among Infants Undergoing Cardiac Surgery: The DECISION Randomized Clinical Trial. JAMA. 2020 Jun 23;323(24):2485-2492. doi: 10.1001/jama.2020.8133. PMID 32573670